CLINICAL TRIAL: NCT06169748
Title: Efficacy of Unihemispheric Concurrent Dual-Site Anodal Transcranial Direct Current Stimulation Combined With Therapeutic Exercise on Pain in Fibromyalgia
Brief Title: UHCDS a-tDCS + TE in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UHCDS a-tDCS+ TE FM Pain
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Neuromodulation; Therapeutic exercise; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real UHCDS a-TDCS + Therapeutic Exercise (Experimental): Real unihemispheric concurrent dual-site anodal transcranial direct current stimulation combined with therapeutic exercise.
  Interventions: Device: Real UHCDS a-tDCS; Device: Therapeutic exercise
- Sham UHCDS a-TDCS + Therapeutic Exercise (Sham Comparator): Sham unihemispheric concurrent dual-site anodal transcranial direct current stimulation combined with therapeutic exercise.
  Interventions: Device: Sham UHCDS a-tDCS; Device: Therapeutic exercise
- Therapeutic Exercise (Active Comparator): Therapeutic Exercise.
  Interventions: Device: Therapeutic exercise

INTERVENTIONS:
Device: Real UHCDS a-tDCS — Real UHCDS a-tDCS (STARTSTIM® 8 stimulator, Neuroelectric Barcelona, Spain) for ten sessions (three sessions per week in weeks 1 and 2; and one session per week in weeks 3, 4, 5 and 6). UHCDS a-tDCS is a galvanic current applied by a cap for 20 minutes at an intensity of 2 milliamps.
  Arms: Real UHCDS a-TDCS + Therapeutic Exercise
Device: Sham UHCDS a-tDCS — Sham UHCDS a-tDCS (STARSTIM® 8 stimulator, Neuroelectric Barcelona, Spain) for ten sessions (three sessions per week in weeks 1 and 2; and one session per week in weeks 3, 4, 5 and 6). Sham tDCS will be applied for the same time than real UHCDS a-tDCS.
  Arms: Sham UHCDS a-TDCS + Therapeutic Exercise
Device: Therapeutic exercise — The therapeutic exercise program will include aerobic exercise and muscle strengthening in the same days as UHCDS a-tDCS. The program will last 30-45 minutes.

SUMMARY:
The present study aims to investigate the effect of a Unihemispheric Concurrent Dual-Site anodal Transcranial Direct Current Stimulation combined with therapeutic exercise on pain in subjects with FM.

DETAILED DESCRIPTION:
Fibromyalgia (FM) syndrome is characterized as a cardinal symptom of chronic pain. It is one of the rheumatic diseases with the greatest impact on quality of life.

Although the etiology and pathophysiology are not yet completely clear, FM is related to specific changes in brain activity, such as a decrease in blood flow in the thalamus, caudate nucleus and pons tegmentum. This could be related to the appearance of a disorder in pain regulation, characterized by an alteration of the sensory and pain process in the central nervous system, due to neuroplastic changes in the neural circuits related to pain. Imaging studies have shown that FM could be associated with functional changes in the brain, such as a reduction in connectivity in efferent pain inhibitory pathways and central sensitization in afferent pain pathways, resulting in an increase in pain perception.

The most common FM treatment guidelines recommend aerobic exercise as the only non-pharmacological therapy with level A recommendation in the treatment of FM. In the same way, it concludes that it is more than recommended to combine therapies assuming synergistic effects between them.

Neuromodulation treatments with transcranial direct current stimulation (tDCS) have been shown to induce significant analgesia in FM through the modification of sensory processing of pain by thalamic inhibitory circuits. To date, the few studies that have combined tDCS and therapeutic exercise in FM have applied tDCS to the primary motor cortex (M1) in isolation. Currently, several studies conclude that Unihemispheric Concurrent Dual-Site anodal Transcranial Direct Current Stimulation (UHCDS a-tDCS) on the dorsolateral prefrontal cortex (DLPFC) and M1 produces a 50% greater modulation of corticospinal excitability in healthy subjects. To date, there is no study that has evaluated the effectiveness of this novel application of tDCS in subjects with FM on pain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Fulfilled the 2010 American Colleague of Rheumatology criteria for fibromyalgia.
* Usual pain intensity of 4 or more points on a visual analogue scale.
* Able to participated in a therapeutic exercise program.
* Understanding of spoken and written Spanish.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Metallic implants in the head.
* Tumor, trauma or surgery in the brain.
* Epilepsy or stroke.
* History of substance abuse in the last 6 months.
* Use of carbamazepine in the last 6 months.
* Diagnosed psychiatric pathology.
* Rheumatic pathology not medically controlled.
* Coexisting autoimmune pathology.
* Chronic inflammatory disease (rheumatoid arthritis, erythematosus systemic lupus, inflammatory bowel disease).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity. | Baseline; inmediately after intervention; 3-months after intervention.
  It will be measured with a visual analog scale (VAS) of 100 millimeters in length. The subject has to indicate the level of pain he feels, being 0 the absence of pain and 100 the maximum imaginable.
Referred pain area after suprathreshold pressure stimulation. | Baseline; inmediately after intervention; 3-months after intervention.
  A pressure algometer (Force Ten™, Wagner Instruments, USA) will be used. It will be performed on the infraspinatus muscle (point equidistant between the midpoint of the spine of the scapula, the inferior angle of the scapula and the midpoint of the medial border of the scapula) at a constant suprathreshold pressure (20% above the pressure pain threshold) for 60 seconds.

SECONDARY OUTCOMES:
Anxiety. | Baseline; inmediately after intervention; 3-months after intervention.
  The version adapted to Spanish from the State Scale (STAI-ES) of the State-Trait Anxiety Inventory (STAI) will be used. STAI-ES ranges from 0 to 60 points, with higher values indicating higher levels of anxiety.
Pain catastrophizing. | Baseline; inmediately after intervention; 3-months after intervention.
  The Spanish version of the Pain Catastrophizing Scale (PCS) will be used. PCS ranges from 0 to 52 points, with higher values indicating higher levels of catastrophizing.
Depression. | Baseline; inmediately after intervention; 3-months after intervention.
  The adaptation to the Spanish of Beck Depression Inventory II (BDI-II) will be used. BDI-II ranges from 0 to 63 points, with higher values indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Arroyo Fernández, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Hospital General Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain